CLINICAL TRIAL: NCT03587298
Title: Use of Shear Wave Elastography in Adolescents and Children With Obesity to Assess Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Use of Shear Wave Elastography to Assess Non-alcoholic Fatty Liver Disease (NAFLD)
Acronym: NAFLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 18-056
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: NAFLD
Keywords: ShearWave Elastography
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: NAFLK criteria met (by definition: sonographic fatty liver)
  Interventions: Procedure: Real-Time (Supersonic)- 2D shear wave elastography (rt-SWE)
- Group 2: Control group: matched age; no NAFKL
  Interventions: Procedure: Real-Time (Supersonic)- 2D shear wave elastography (rt-SWE)

INTERVENTIONS:
Procedure: Real-Time (Supersonic)- 2D shear wave elastography (rt-SWE) — The SWE is carried out intercostally. If possible, the patient should hold the breath for 5-10 seconds. So-called colour charts are used, which indicate the derived liver stiffness in colour-coded form. In addition to the visual assessment of these colour charts, the quantitative ROI-based measurement of the SWE in kPa is performed in the "hardest" appearing areas. The measurement is performed at 5 different sites of the liver parenchyma and all SWE values are recorded.

SUMMARY:
The aim of this study is to test a non-invasive imaging technique to reliably diagnose NAFLD in children and adolescents with obesity and assess the degree of fibrosis.

DETAILED DESCRIPTION:
NAFLD (non-alcoholic fatty liver disease) is by far the most common form of chronic liver disease worldwide. It is estimated that it affects up to 1/3 of the adult population in industrialized countries and additionally more and more children are affected. The term NAFLD covers a broad spectrum of diseases ranging from simple hepatic steatosis (accumulation of fat in hepatocytes) to NASH (non-alcoholic steatohepatitis). The latter is a progression of liver steatosis with inflammation, fibrosis and chronic inflammatory structural changes. Up to 20% of a NASH develops liver cirrhosis, more rarely also a hepatocellular carcinoma.

It is known that the degree of fibrosis is the most important parameter for the clinical course and prognosis. In addition, patients with mild lobular inflammation or fibrosis (regardless of severity) have an increased risk of developing NASH compared to patients with exclusive steatosis. A significant number of patients with NAFL may develop fibrotising NASH (5-20%). This is particularly the case when metabolic factors continue to deteriorate.

Liver biopsy remains the gold standard for the diagnosis of NAFLD. In particular, differentiation between NAFL and NASH and the degree of fibrosis are still only possible using histology. The invasive nature of the procedure involves risks to the patient's health such as bleeding, injuries to other organs or nerves, and complications of anesthesia. Furthermore, since the biopsy is taken selectively as a liver biopsy, it is possible to test a sample that does not adequately represent the degree of actual fibrosis, since regional differences in the severity of liver fibrosis can often be present. In addition, the liver biopsy is associated with considerable costs. Accordingly, liver biopsy is not an optimal diagnostic procedure and is hardly suitable as a diagnostic method for short-term follow-up under therapy. For this reason, a reliable, non-invasive method has long been sought to diagnose NAFLD, to distinguish NASH from steatosis, to assess the degree of fibrosis and which allows a less stressful assessment of the course of the liver.

Imaging procedures are available here. B-image sonography is already routinely used in children and adolescents with suspected or proven NASH for the detection of liver remodeling processes, in particular fibrosis. B-scan sonography is an excellent method for determining the presence and extent of hepatic steatosis, but the detection and graduation of liver fibrosis using B-mode sonography is only possible in very advanced stages.

In recent years, the determination of tissue stiffness in various organ systems and their pathologies, such as the breast, tendons and liver, has been successfully used in adults. Individual reports in adults give first indications that liver remodelling processes, in particular fibrosis by means of shear wave elastography (SWE), can be diagnosed in early stages. However, the evidence of the use of SWE in children to assess liver parenchyma changes, especially in NAFLD, is still insufficient. Therefore, in this study it will be investigated whether the rt-SWE provides reproducible values for liver stiffness and fibrosis in children and adolescents and by that a reliably diagnosis of NAFLD and assessment of the degree of fibrosis is possible.

The planned clinical examination and blood collection for laboratory chemical examinations are part of the routine follow-up of patients with obesity and steatosis hepatis. There will be no additional examinations, so there will be no greater burden on the young patients and no additional time expenditure.

ELIGIBILITY:
Inclusion Criteria:

* male and male children and adolescents aged 6-18 years
* obesity with a BMI above percentile 95 according to Kromeyer-Hauschild
* NAFLD criteria met (by definition: sonographic fatty liver)
* written informed consent
* patients of matching age are included in the control group without any indication of NAFLD

Exclusion Criteria:

* other chronic liver diseases
* alcohol consumption (more than 20g for girls and 30g for boys per day), after explicit anamnesis
* persons who are accommodated in an institution by court or official order

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The patient group is recruited from the obesity consultation hour as well as the emergency consultation hour and the wards of the Clinic for Paediatrics and Youth Medicine at the University Hospital Aachen.
  The control group is recruited from the group of outpatients and inpatients receiving abdominal sonography from another indication and show no sonographic or laboratory chemical evidence of NAFLD. Patients in the control group are evaluated once.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Assess non-alcoholic fatty liver disease in adolescents and children with obesity by use of shear wave elastography | 12 month
  stiffness (in kilopascals) of the liver measured with real-time shear wave elastography (RT-SWE) and hence regarding the amount of fibrosis in chronic liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Angeliki Pappas, Dr. med., Principal Investigator — Paediatric Clinic; RWTH Aachen University Hospital
Locations (1):
- Paediatric Clini; RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany